CLINICAL TRIAL: NCT04369066
Title: COVID-19 Study of the Serological Response Against the SARS-CoV-2 Virus in 2 Types of Employees, Hospital and Non-hospital, at Institute Curie and Institute Pasteur
Brief Title: COVID-19 Study of the Serological Response Against the Severe Acute Respiratory Syndrome (SARS) Coronavirus 2 (CoV-2) Virus in 2 Types of Employees, Hospital and Non-hospital, at Institute Curie and Institute Pasteur
Acronym: Curie-O-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IC 2020-07
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2023-11

CONDITIONS: Volunteers From the Institute Curie and Institute Pasteur Staff Who Are Not Showing Active SARS-CoV-2 Infection
Keywords: Adults; Volunteers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects who are not showing active SARS-Cov2 infection (Other)
  Interventions: Diagnostic Test: Blood samples (collection of 5 mL of blood in a dry tube); Diagnostic Test: Nasopharyngeal swabs

INTERVENTIONS:
Diagnostic Test: Blood samples (collection of 5 mL of blood in a dry tube) — A nurse will take blood samples under safe conditions compatible with the pandemic period and while respecting the protection of the volunteer's personal data.
  The blood samples will be taken at 4 times for Institute Curie and Institute Pasteur: T0, between 6 weeks and 3 months ,6 months and 12 months post-inclusion.
  For volunteers already included at Institute Curie : in case of proved (RT-PCR+ or antigenic +) or very likely (anosmia and/or ageusia, and/or digestive syndrome with associated respiratory signs) between 2 sampling times already planned in the flow chart, blood samples shall be performed, if time since last planned sampling(s) has been more than 3 weeks or if time until next sampling(s) is more than 3 weeks.
  The serum samples will be extracted and collected prospectively from the blood samples.
  For each blood sample, a sample number will be assigned by the laboratory management system of the Department of Biology at Institut Curie.
Diagnostic Test: Nasopharyngeal swabs — The nasopharyngeal swabs will be performed between 6 weeks and 3 months, 6 months and 12 months post-inclusion for Institute Curie staff with at least one of the following criteria: have had RT-PCR+, and/or presence of antibodies at the 95% threshold, and/or anosmia/ageusia, and/or digestive syndrome with associated respiratory signs.
  The nasopharyngeal swab shall also be proposed to volunteers not meeting the above listed criteria to have a control group (about 100 volunteers).
  For volunteers already included at Institute Curie : in case of proved (RT-PCR+ or antigenic +) or very likely (anosmia and/or ageusia, and/or digestive syndrome with associated respiratory signs) infection between 2 sampling times, nasopharyngeal swabs shall be performed if time since last planned sampling(s) has been more than 3 weeks or if time until next sampling(s) is more than 3 weeks.
  The nasopharyngeal swabs will be performed at T0 for Institute Pasteur staff so 4 times in total.

SUMMARY:
This research proposes to study a large healthy population active for the presence of antibodies directed against the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) virus and this over time.

After verification of the inclusion criteria and information by the coordinating investigative doctor, the volunteers sign a written consent. A nurse will take blood samples under safe conditions compatible with the pandemic period and while respecting the protection of the volunteer's personal data.

The blood samples will be taken at 4 times for Institute Curie and Institute Pasteur: T0 (day of inclusion), between 6 weeks and 3 months ,6 months and 12 months post-inclusion.

Each blood sample consists of a collection of 5 mL of blood in a dry tube. The serum samples will be extracted and collected prospectively from the blood samples.

The nasopharyngeal swabs will be performed at 3 times: , between 6 weeks and 3 months, 6 months and 12 months post-inclusion for Institute Curie staff who have had at least one of the following four criteria on the sample or questionnaire carried out at T0:

* have had RT-PCR+
* and/or presence of antibodies at the 95% threshold
* and/or anosmia/ageusia
* and/or digestive syndrome with associated respiratory signs. In case of infection between sampling times, if the volunteer meets one of the four criteria above, a nasopharyngeal swab will be performed during the following visits.

The nasopharyngeal swab shall also be proposed to volunteers not meeting the 4 above listed criteria in order to have a control group (about 100 volunteers) for future statistical analyses.

If the volunteers accept, naso-pharyngeal swab shall be performed between 6 weeks and 3 months, 6 months and 12 months after inclusion.

For volunteers already included at Institute Curie : in case of proved (RT-PCR+ or antigenic +) or very likely (anosmia and/or ageusia, and/or digestive syndrome with associated respiratory signs) between 2 sampling times already planned in the flow chart, blood samples and nasopharyngeal swabs shall be performed.

Those shall be performed if time since last planned sampling(s) has been more than 3 weeks or if time until next sampling(s) is more than 3 weeks.

The blood samplings and nasopharyngeal swabs will be performed at 4 times for Institute Pasteur personnel: at T0 (inclusion day), between 6 weeks and 3 months, at 6 months and 12 months post-inclusion

ELIGIBILITY:
Inclusion Criteria:

1. Person, adult volunteer outside of any acute infectious episode with SARS-CoV-2* (see paragraph indication), working at the Institute Curie and able to exercise their professional activity on one of the 3 sites of the Institute Curie: Paris, Orsay or Saint Cloud, or on the Campus of the Institute Pasteur.
2. Person aged 18 or over.
3. Information and consent of the person to the procedures related to the study (cf. information note / consent).

From November 2020, person having presented at least one of the following criteria since January 2020:

* A positive diagnostic test for SARS-COV-2 by PCR on a nasopharyngeal sample or antigenic test,
* A positive SARS-CoV-2 serology,
* An anosmia or / and an ageusia,
* A respiratory infection ** associated with digestive signs **

whatever the working methods during confinement * Subjects who are not showing active SARS-CoV-2 infection are considered volunteers at the time of inclusion: people with no clinical signs ** suggestive of SARS-CoV-2 infection at the time of collection or having had an end of symptoms for more than 7 days [1].

** fever, fatigue, cough, shortness of breath, difficulty to breath, loss of taste or smell, headache, body aches, conjunctivitis or cold, digestive problems (vomiting, diarrhea), whether or not the signs led to sick leave, treatment and / or hospitalization [2].

Exclusion Criteria:

* Declaration by the subject of signs suggestive of Coronavirus Infectious Disease 2019 (COVID-19) infection with SARS-CoV-2 in progress or for which the end of symptoms dates from less than 7 days
* Inability to submit to study monitoring for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1971 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Antibodies against the SARS-CoV-2 virus in serum at inclusion | 1 day
  Detection of antibodies against the SARS-CoV-2 virus with serological tests
Antibodies against the SARS-CoV-2 virus in serum at 1 month | 1 month
  Detection of antibodies against the SARS-CoV-2 virus with serological tests
Antibodies against the SARS-CoV-2 virus in serum at 3 months | 3 months
  Detection of antibodies against the SARS-CoV-2 virus with serological tests
Antibodies against the SARS-CoV-2 virus in serum at 6 months | 6 months
  Detection of antibodies against the SARS-CoV-2 virus with serological tests
Antibodies against the SARS-CoV-2 virus in serum at 12 months | 12 months
  Detection of antibodies against the SARS-CoV-2 virus with serological tests

SECONDARY OUTCOMES:
Comparative performance of anti-SARS-CoV-2 antibody detection techniques | 9 months
  Comparative performance of anti-SARS-CoV-2 antibody detection techniques (sensitivity and specificity of serological tests)
Prevalence of immune subjects for SARS-CoV-2 | 3 months
  Prevalence of immune subjects for SARS-CoV-2 in a well-defined active healthy population, working at the hospital or not, leading to variable exposure levels
Nature and quantity of anti-SARS-CoV-2 antibodies | 3 months
  Nature and quantity of anti-SARS-CoV-2 antibodies: ImmunoglobulinM, ImmunoglobulinG and ImmunoglobulinA)
Evolution of the different antibodies against the SARS-CoV-2 virus over time. | 6 months
  The analysis of the evolution of serology results over time will be done by a mixed model taking into account the repeated framework of the data of a subject
Prevalence of Anti-covid IgA response in the nasal mucosa | 6 months
  Prevalence of Anti-covid IgA in volonteers RT/PCR+ and/or presence of antibodies at the 95 % threshold and/or COVID symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, PhD, Study Director — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Background] Anna F, Goyard S, Lalanne AI, Nevo F, Gransagne M, Souque P, Louis D, Gillon V, Turbiez I, Bidard FC, Gobillion A, Savignoni A, Guillot-Delost M, Dejardin F, Dufour E, Petres S, Richard-Le Goff O, Choucha Z, Helynck O, Janin YL, Escriou N, Charneau P, Perez F, Rose T, Lantz O. High seroprevalence but short-lived immune response to SARS-CoV-2 infection in Paris. Eur J Immunol. 2021 Jan;51(1):180-190. doi: 10.1002/eji.202049058. Epub 2020 Dec 23. PMID 33259646